CLINICAL TRIAL: NCT06638749
Title: Effect of Tranexamic Acid on Blood Loss in Reverse Total Shoulder Arthroplasty
Brief Title: Effect of TXA on Blood Loss in Reverse Total Shoulder Arthroplasty
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Administrative withdrawal-study not approved by IRB
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00142552
Record Dates: First submitted 2019-04-24; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2019-04

CONDITIONS: Shoulder Arthritis; Blood Loss, Surgical; Tranexamic Acid Adverse Reaction
MeSH Terms: conditions — Blood Loss, Surgical | interventions — Tranexamic Acid; Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding tables to be held by investigational pharmacy. Surgeon and patient will be blinded from administration of TXA versus saline placebo.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tranexamic acid (Experimental): The experimental group will receive 1 gram of intravenous tranexamic acid at skin incisions and 1 gram at skin closure.
  Interventions: Drug: Tranexamic Acid
- Normal Saline (Placebo Comparator): The control group will receive 100 ml of normal saline, 50 ml at incision and 50 ml at closure instead of tranexamic acid.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Tranexamic Acid — Administration of tranexamic acid
  Arms: Tranexamic acid
Drug: Normal Saline — Administration of normal saline
  Arms: Normal Saline

SUMMARY:
Tranexamic acid (TXA) is a synthetic anti-fibrinolytic agent that has been well studied and routinely used for hip and knee arthroplasty. In hip and knee arthroplasty, the use of tranexamic acid decreases blood loss and the need for transfusion without increasing the risk of thromboembolic events. Due to the increased use of reverse total shoulder arthroplasty in the treatment of shoulder pathology, there has been interest in making the procedure safer for patients. TXA is a promising drug which could be useful to surgeons as they seek to achieve this goal, however, it has not been extensively studied in this setting. The purpose of this prospective randomized, controlled study is to determine the effectiveness and safety of using tranexamic acid to decrease blood loss in reverse total shoulder arthroplasty.

DETAILED DESCRIPTION:
Study Title: Effect of TXA on intra-operative blood loss in reverse total shoulder arthroplasty, a randomized controlled trial I. Purpose, Background and Rationale A. Aim and Hypotheses 1. Tranexamic acid (TXA) is a synthetic anti-fibrinolytic agent that has been well studied and routinely used for hip and knee arthroplasty. In hip and knee arthroplasty, the use of tranexamic acid decreases blood loss and the need for transfusion without increasing the risk of thromboembolic events. Due to the increased use of reverse total shoulder arthroplasty in the treatment of shoulder pathology, there has been interest in making the procedure safer for patients. TXA is a promising drug which could be useful to surgeons as they seek to achieve this goal, however, it has not been extensively studied in this setting. The purpose of this prospective randomized, controlled study is to determine the effectiveness and safety of using tranexamic acid to decrease blood loss in reverse total shoulder arthroplasty. 2. Investigators hypothesize that patients who receive an intra-operative administration of tranexamic acid (TXA), as compared to control patients who do not receive TXA, will:

1. Have decreased intra-operative blood loss as estimated by the operating surgeon
2. Have a smaller drop in hemoglobin as measured with a complete blood count performed on post-op day one
3. Have less post-operative drain output
4. Have no increase in the rate of adverse events including venous thromboembolic events or infection. B. Background and Significance Tranexamic acid (TXA) is a synthetic lysine analog which competitively inhibits the activation of plasminogen to plasmin, preventing the breakdown of the fibrin matrix. This effectively stabilizes clot formation and has been shown to decrease blood loss in multiple settings. In total hip and total knee arthroplasty, the use of TXA has been shown to decrease blood loss and the need for blood transfusion in the perioperative period.

Despite its clot-stabilizing effect, TXA has not been shown to increase the risk of thromboembolic events (Duncan et al.,2015; Yang et al., 2013). Intravenous tranexamic acid is FDA approved for use in hemophilia and to reduce bleeding complications for The use of TXA in total shoulder arthroplasty has been less well studied. The rate of blood transfusion in these procedures, although lower than hip and knee arthroplasty, is reported between 4 and 43%. A retrospective study by Hardy et al. in 2013 showed an overall transfusion rate of 7.4%, with intra-operative estimated blood loss being an independent risk factor for transfusion. The risks associated with blood transfusion have been decreased with modern screening methods, however, there are multiple studies specific to hip and knee arthroplasty showing an association with adverse events such as infection, venous thromboembolic events, and even mortality. In addition, Grier et al.

used the Medicare Standard Analytic files database to study over 7500 patients who received a blood transfusion after anatomic or reverse total shoulder arthroplasty and compared them to age- and gender-matched controls. They found a statistically increased rate of myocardial infarction, pneumonia, sepsis, and cerebrovascular accident in the transfusion group. Methods to reduce blood loss and, therefore, the rate of transfusion are clearly invaluable in improving patient outcomes for shoulder arthroplasty. A few studies over the last two years have looked at the role of tranexamic acid in total shoulder arthroplasty. Two retrospective review studies have shown that TXA can be effective in decreasing blood loss and length of hospital stay in patients undergoing reverse or anatomic total shoulder arthroplasty (Abilgaard et al., 2016; Friedman et al., 2018). A randomized control trial including 54 patients undergoing reverse or anatomic total shoulder arthroplasty demonstrated decrease blood loss, patient-reported pain, and hematoma formation (Pauzenberger et al., 2017). One study specific to reverse total shoulder arthroplasty showed a decrease in blood loss (1124 ml in the control group, 411 in the TXA group). In this study, 7 transfusions were reported in the control group compared to 3 in the TXA group. The patients in this study received prophylactic heparin during their hospital stay. A meta-analysis of 5 studies, including those described above, included a total of 629 patients and showed that patients receiving TXA had decreased blood loss. There was no increase in adverse events in the TXA group patients. These studies indicate that tranexamic acid may be effective in decreasing the amount of blood loss during reverse total shoulder arthroplasty. However, these studies are heterogeneous in that several of them include patients undergoing either reverse or anatomic total shoulder arthroplasty, which are inherently different procedures regarding the implants used and the specific risks involved. Please see the literature cited section for full citations. C. Rationale This study aims to add to the currently small body of literature regarding the role of tranexamic acid in reverse total shoulder arthroplasty. Several elements of our study are unique. First, investigators will include only patient's undergoing reverse total shoulder arthroplasty. In addition, patients will not receive chemoprophylaxis against deep venous thrombosis. This is the standard of care at our institution, where it has been noted less blood loss and a decreased transfusion rate as compared to the published studies.

II. Research Plan and Design

A. Study Objectives:

1. Determine whether the use of tranexamic acid decreases intra-operative blood loss, postoperative change in hemoglobin, and amount of post-operative drain output in reverse total shoulder arthroplasty.
2. Determine whether the use of tranexamic acid effects the rate of adverse events including thromboembolic events, infection, and hematoma. III. Study Type and Design: Prospective randomized controlled trial. IV. Sample size, statistical methods, and power calculation

1. Investigators will perform randomization in a 1:1 ratio between the control and TXA groups. The plan is to perform a t-test to analyze normal data and Mann-Whitney-rank sum test to analyze non-normal data. This applies to the quantitative data that will be collected: estimated blood loss, change in hemoglobin, and drain output. Chi squared analysis will be used to analyze data that is categorical such as transfusion, hematoma, and adverse events. 2. Blinding will be performed and controlled by the pharmacy. The code to the blind will be maintained by pharmacy. In the event of an adverse event or unforeseen complication during or after the procedure, the anesthesiology or operative team will be able to break the code to direct treatment by communicating with the pharmacy. 3. Based on the published results and our typical estimated blood loss, investigators estimate an average blood loss of 150 ml in the TXA group and 250 +/- 100 ml for the control group.

With a p value of 0.05, 16 patients will need to be enrolled in each group to have a study with adequate power. A maximum of 60 patients will be enrolled per group. No pilot testing will be performed.

V. Subject Criteria (See Vulnerable Populations appendix, if applicable):

1. Inclusion criteria: Plan to include patients undergoing primary reverse total shoulder arthroplasty regardless of age and gender.
2. Exclusion criteria: Exclusion criteria will include patients on anticoagulation at the time they are scheduled for surgery. There will be additional exclusion of patients with known clotting or bleeding abnormalities.
3. Withdrawal/Termination criteria: Adverse events as detailed above.
4. Patients may participate in other studies while participating in this study. E. Specific methods and techniques used throughout the study

1. Laboratory tests: Pre and post-operative complete blood counts (CBC). Pre-operative CBCs are routinely obtained at the pre-anesthesia testing visit. Post-operative CBC on post-operative day one is standard of care at our institution. 2. Study Procedures: Reverse total shoulder arthroplasty will be performed as scheduled by the operating surgeon. Regardless of participation in the study, this will be performed through a standard deltopectoral approach. Cases are usually scheduled for 2-3 hours.

3. As stated above, the complete blood counts, recording of drain output, estimation of surgical blood loss and documenting transfusions are all part of usual standard therapy.

The surgical procedure will also be performed in the usual manner. 4. Samples obtained will be handled per hospital protocol and sent to the hospital laboratory for analysis and disposal. 5. Patients will be approached in the orthopedic clinic after they have been scheduled for reverse total shoulder arthroplasty. The project will be explained to each patient and they will be given the opportunity to enroll if they choose. Informed consent will be obtained at that time. Randomization will be performed in a 1:1 ratio between the control and TXA groups. Blinding will be performed by the investigational pharmacy, which will maintain the blinding tables. The staff anesthesiologist involved in the procedure will be able to break the blind for patient safety reasons if necessitated by the clinical scenario intraoperatively.

The procedure will be completed in the standard manner. Intra-operative blood loss will be estimated by the performing surgeon, Dr. Tyler Fox. Hemoglobin values will be recorded pre-operatively at the patient's pre-anesthesia testing visit and compared to the value on post-operative day one. In addition, drain output will be measured on the first post-operative day. Adverse events such as hematoma, venous thromboembolic events, and adverse events requiring hospitalization will be monitored until the patient's second post-operative follow up visit (6-8 weeks post-operatively). Investigators will record all transfusions in the post-operative period. Statistical analysis will be performed while the group identities are blinded to the investigator. Normal data will be analyzed with a t-test and non-normal data will be analyzed with the Mann-Whitney rank U test. This applies to quantitative data such as estimated blood loss, change in hemoglobin, and drain output. Categorical data such as need for transfusion, hematoma, and adverse events will be analyzed with Chi squared analysis. F. Risk/benefit assessment

1. Physical risk Study arm patients will have the risks associated with administration of TXA. Previous studies have shown that administration of TXA is well tolerated and does not increase the risk of significant adverse events. There has been no reported increase in venous thromboembolic events in arthroplasty patients. Please see above literature review. Side effects do include nausea, vomiting, diarrhea, and headaches which patients will be treated for symptomatically during their admission. Control patient's will have their procedure as planned and will be exposed to minimal additional risk from the administration of normal saline.
2. Psychological risk N/A
3. Social risk N/A
4. Economic risk N/A
5. Potential benefit of participating in the study

   1. Benefits to patient: Study arm patients will potentially receive the benefit of decrease in peri-operative blood loss if our results are similar to previous studies.
   2. Benefits to patient's population: Reverse total shoulder arthroplasty is a successful procedure any becoming more widespread. This study could benefit patients undergoing reverse total shoulder arthroplasty.
   3. Benefits to society: Reduction in complications and blood transfusions could improve the efficiency of healthcare delivered. G. Location where study will be performed: KU Medical Center

ELIGIBILITY:
Inclusion Criteria:

* Candidate for reverse total shoulder arthroplasty

Exclusion Criteria:

* Patient's on anti-coagulation at the time they are scheduled for surgery will be excluded from participation. In addition, patients with known clotting or bleeding abnormalities will be excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-05-01 (Estimated); Primary Completion 2020-12-01 (Estimated); Study Completion 2024-10-10 (Actual)

PRIMARY OUTCOMES:
Intra-operative blood loss | At time of surgery
  Estimated by operating surgeon

SECONDARY OUTCOMES:
Drain output | Post operative day one
  Recorded on post operative day 1
Change in hemoglobin | Pre- versus post-operatively
  Between pre-operative and post-operative CBC values
Adverse events | For 6-8 weeks post operatively
  transfusion, hematoma, venous thromboembolic events, and adverse events requiring hospitalization will be monitored until the patient's second post-operative follow up visit (6-8 weeks post-operatively).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No